CLINICAL TRIAL: NCT03005197
Title: A Prospective Study to Assess the Diagnostic Accuracy of Laser Doppler Flowmetry in Assessing Pulp Vitality of Traumatised Teeth in Paediatric Patients
Brief Title: Laser Doppler Flowmetry in Assessing the Vitality of Traumatised Teeth
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Leeds (Other)
Responsible Party: Principal Investigator, Nahar Ghouth, Principal Investogator, University of Leeds
Other Study IDs: 1
Record Dates: First submitted 2016-12-22; First posted 2016-12-29 (Estimated); Last update posted 2017-01-05 (Estimated); Status verified 2017-01

CONDITIONS: Dental Trauma
MeSH Terms: interventions — Laser-Doppler Flowmetry

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Laser Doppler Flowmetry
  Other Names: LDF

SUMMARY:
Teeth injuries are considered one of the most challenging events that occur in dentistry, especially in children. After an injury, there is a possibility that the blood supply to the tooth may become affected and compromised leading to nerve and blood vessels death with the tooth described as a non-vital tooth.

The conventional diagnostic tools available to assess tooth nerve/blood supply are not always reliable. Child cooperation and understanding contribute greatly to this shortfall. Failure to assess the vitality of the tooth may result in pain, swelling or infection of the tooth or de-vitalising a normal tooth which may render the tooth weak for the future and possibly losing the tooth.

The laser Doppler flowmetry is a non-invasive, non-painful technique and shown to be more reliable than the traditional techniques. We aim to assess if this device can predict and assess whether the tooth is alive or dead during the follow up visits of the injury along the other conventional tests.

DETAILED DESCRIPTION:
A clinical study will be carried out which consists of a one year follow up to monitoring traumatised front teeth in children attending the department of paediatric dentistry.

The vitality/sensibility of traumatised teeth will be assessed using laser Doppler flowmetry, electrical pulp testing and ethyl chloride. Measurements will be performed by a single operator (chief investigator) and will be carried out at baseline, 3, 6, 9 and 12 months follow up period.

ELIGIBILITY:
Children would be recruited into this study when they:

* Between 6-16 years old.
* Medically fit (ASA I, II).
* Able to communicate using English language.
* Have an acceptable level of cooperation.
* Have at least one traumatised anterior tooth, regardless of the type of trauma, with uncertain pulpal vitality requiring monitoring for a minimum of 12 months and minimal coronal restoration (covering less than half the labial crown surface).
* Have at least one vital and non-traumatised anterior tooth to act as a control.

Exclusion Criteria:

* Medically and mentally compromised children.
* Children with learning disabilities.
* Children with communication barrier including those unable to communicate using English language.
* Heavily restored teeth covering more than half the labial surface of teeth.
* Patients on routine analgesics, antidepressants or antihypertensive drugs.
* Vital teeth with pulp canal obliteration.

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Patients attending the children's dentistry department at Leeds Dental Institute will be assessed for suitability in taking part into this study according to the study inclusion and exclusion criteria.
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2017-02; Primary Completion 2018-05 (Estimated); Study Completion 2018-05 (Estimated)

PRIMARY OUTCOMES:
Sensitivity | One year follow up
Specificity | One year follow up

CONTACTS AND LOCATIONS:
Overall Officials: Nahar Ghouth, Principal Investigator — University of Leeds

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jafarzadeh H. Laser Doppler flowmetry in endodontics: a review. Int Endod J. 2009 Jun;42(6):476-90. doi: 10.1111/j.1365-2591.2009.01548.x. PMID 19459999